CLINICAL TRIAL: NCT05512416
Title: Neoadjuvant Dalpiciclib Plus Letrozole for HR+/HER2- Breast Cancer: A Single Arm, Open Label, Phase II Trial
Brief Title: Neoadjuvant Dalpiciclib Plus Letrozole for HR+/HER2- Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-Ⅱ-040
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; CDK4/6 inhibitor; endocrine therapy; hormone receptor-positive; dalpiciclib; letrozole
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib; Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohort 1 (Experimental): patients with stage IIB-III HR+/HER2- breast cancer
  Interventions: Drug: dalpiciclib plus letrozole

INTERVENTIONS:
Drug: dalpiciclib plus letrozole — Six 4-week cycles of dalpiciclib orally, 150mg, day 1-21, and letrozole orally, 2.5 mg, day 1-28
  Other Names: D+L

SUMMARY:
In this single arm, open label, phase 2 trial, operable patients with stage IIB-III HR+/HER2- breast cancer will be enrolled and receive six cycles of adjuvant dalpiciclib plus letrozole. This study aims to assessed the biological effects and safety of dalpiciclib in combination with letrozole for HR+/HER2- breast cancer in the neoadjuvant setting.

DETAILED DESCRIPTION:
This is a single arm, open label, phase 2 trial aimed to investigate the biological effects and safety of neoadjuvant dalpiciclib in combination with letrozole for HR+/HER2- breast cancer. A total of 35 patients with stage IIB-III HR+/HER2- breast cancer will be enrolled. Six 4-week cycles of adjuvant therapy will be administrated. In each cycle, patients use dalpiciclib orally, 150mg, day 1-21, and letrozole orally, 2.5 mg, day 1-28. Premenopausal or perimenopausal patients should combine ovarian function suppression, including bilateral oophorectomy or treatment with gonadotropin-releasing hormone agonists. The primary endpoint is complete cell-cycle arrest at C1D15, defined as ki67≤2.7%. The secondary endpoints include residual cancer burden, overall response rate, change in Ki67 from baseline to 2 weeks of treatment, preoperative endocrine prognostic index, pathologic complete response, breast-conserving surgery rate and safety profile.

ELIGIBILITY:
Inclusion Criteria： Postmenopausal, premenopausal or perimenopausal women aged ≥18. Postmenopausal was defined as: 1) received bilateral oophorectomy, or aged ≥60; 2) aged <60, reached natural menopause (defined as no menses for 12 or more consecutive months with no other reason for the amenorrhea), and with postmenopausal E2 and FSH level; 3) premenopausal or perimenopausal women may also be enrolled as long as they are willing to receive LHRH agonist therapy during the study； Operable patients with ER+ (>10%), HER2- invasive breast carcinomas, regardless of PR level. HER2- was defined as IHC score of 0+, or IHC score of 2+ with negative ISH (amplification ratio <2.0) according to 2018 ASCO-CAP guideline； Untreated patients with stage IIB-III according to AJCC criteria (8th edition)； Without known hypersensitivity to the study drug or its excipients； A ECOG PS score of 0-1； With the ability to swallow the study drug； With sufficient organ function, including 1) bone marrow function: ANC ≥ 1.5 x 109/L (without growth factors within 14 days); PLT ≥ 100 x 109/L (without corrective therapy within 7 days); Hb ≥ 100 g/L (without corrective therapy within 7 days); 2）liver and kidney function: TBIL ≤ ULN; ALT and AST ≤ 3 × ULN (ALT and AST ≤ 5 × ULN for those with liver metastases); BUN and Cr ≤ 1.5×ULN, and creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula); 3) QT interval ≤ 480 ms from the 12-lead electrocardiogram； Able to undergo all puncture biopsies required by the protocol； Volunteered to participate in this study; signed informed consent; with good compliance and willingness to follow-up；

Exclusion Criteria： Previously treated patients, including chemotherapy, radiotherapy, targeted therapy or endocrine therapy, etc.； Concurrently receiving any anti-tumor treatments other than that prescribed by the protocol； Patients with bilateral breast cancer, inflammatory breast cancer or occult breast cancer； Patients with stage IV breast cancer； Patients with severe liver, kidney, or heart dysfunction； Inability to swallow, with chronic diarrhea, with intestinal obstruction, or with other factors affecting drug administration and absorption； Participated in other clinical trials within 4 weeks before enrollment； Known hypersensitivity to the study drug or its excipients; history of ；immunodeficiency, including HIV positive, HCV positive, active viral hepatitis B, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation； History of any cardiac disease, including: 1) arrhythmias requiring drug treatment or of clinical significance; 2) myocardial infarction; 3) heart failure; 4) any other cardiac disease to be inappropriate for this trial judged by the investigator； Women who are pregnant or breastfeeding, women of childbearing potential who test positive for pregnancy test at baseline, or women of childbearing potential who are unwilling to use effective contraception during the study； With serious concomitant disease that endanger safety, or interferes with the ability to complete the study judged by the investigator (including, but not limited to, uncontrolled hypertension, severe diabetes, active infection, etc.)； History of neurological or psychiatric disorders, including epilepsy or dementia; or any other condition inappropriate for this study deemed by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Complete cell-cycle arrest at C1D15, defined as ki67≤2.7% | up 2 years
  From the date into this study(signed ICF) to C1D15,defined as ki67≤2.7%

SECONDARY OUTCOMES:
residual cancer burden | up 2 years
  The percentage of residual tumors after neoadjuvant therapy is assessed according to breast tumor bed tumors and regional lymph nodes
objective response rate | up 2 years
  The rate of CR and PR,determined using RECIST v1.1 criteria
change in Ki67 from baseline to 2 weeks of treatment | up 2 years
  change in Ki67 from baseline（From the date into this study(signed ICF) ） to 2 weeks of treatment
preoperative endocrine prognostic index | up 2 years
  Prognostic indicators of preoperative endocrine therapy, including mass size after neoadjuvant endocrine therapy, lymph node status, ki67 levels, and estrogen receptor (ER) status
pathologic complete response | up 2 years
  After neoadjuvant therapy, there are no residual invasive tumors in the primary focus and regional lymph nodes of breast cancer, but ductal carcinoma in situ may be present(ypT0/is ypN0)
breast-conserving surgery rate | up 2 years
  The number of cases that actually underwent breast-conserving surgery after surgery accounted for the percentage of all breast cancer patients who underwent surgery
safety profile | up 2 years
  Adverse events (AE) and severe adverse events (SAEs) are recorded. Refer to NCI-CTC AE 5.0 standard